CLINICAL TRIAL: NCT01350193
Title: Manuka Honey Irrigation After Endoscopic Sinus Surgery
Brief Title: Manuka Honey Irrigation After Sinus Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, MD FRCSC FARS, Principal Investigator, Director of St Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHI-2011
Record Dates: First submitted 2011-05-03; First posted 2011-05-09 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Sinusitis
Keywords: Manuka Honey; Irrigation; Endoscopic Sinus Surgery
MeSH Terms: conditions — Sinusitis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Nasal Irrigation (Active Comparator): Saline Nasal Irrigation is actively being used as the standard of care. It does not contain any active ingredients.
  Interventions: Other: Saline Irrigation
- Manuka Honey Irrigation (Experimental): Manuka Honey Irrigation involves the experimental treatment of manuka honey nasal irrigation.
  Interventions: Device: Manuka Honey

INTERVENTIONS:
Device: Manuka Honey — The use of the nasal irrigation on post-operative day #1. 30mL of the nasal irrigation will be applied to each nostril by a 60mL Toomey syringe (given to patient at pre-operative clinic visit) twice a day (once in am, once in pm). This will continue until the 6 month post-op visit.
  Other Names: Irrigation; Endoscopic Sinus Surgery
  Arms: Manuka Honey Irrigation
Other: Saline Irrigation — The use of the nasal irrigation on post-operative day #1. 30mL of the nasal irrigation will be applied to each nostril by a 60mL Toomey syringe (given to patient at pre-operative clinic visit) twice a day (once in am, once in pm). This will continue until the 6 month post-op visit.
  Other Names: Control; Endoscopic Sinus Surgery
  Arms: Saline Nasal Irrigation

SUMMARY:
All adult (over 19 years) patients undergoing sinus surgery for chronic rhinosinusitis (CRS) or allergic fungal sinusitis (AFS) that do not meet the exclusion criteria will be included in the study.

All participants enrolled in the study will receive antibiotic (Clavulin) therapy 1-week pre-and post-operatively and oral steroid therapy 1-week pre-operatively and post-operatively.

Randomization of patients to the Manuka Honey irrigation (treatment arm) and Saline irrigation (standard of care) will occur on the day of surgery.

Participants in both study arms will undergo the standard post-operative endoscopic sinus surgery follow-up. This includes follow-up appointments at 6 days, 5 weeks, 3 months, and 6 months of the post-operative period. During these appointments, the surgeon will assess the post-operative appearance (Philpott-Javer Sinus Rating System), number of infections, pain, and 1st week post-operative bleeding (only at 6 day visit).

The Sino-Nasal Outcome Test (SNOT-22) questionnaire is to be completed by the study participants at 6 days, 5 weeks, and 3 months of the post-operative period. The SNOT-22 is a 5-minute questionnaire consisting of 22 questions, which asks participants to rate their sinus symptoms and social/emotional consequences of their nasal disorder from "no problem" to "problem as bad as it can be."

DETAILED DESCRIPTION:
All patients in this study will undergo endoscopic sinus surgery. This is the mainstay of treatment for patients with refractory sinus disease.

All patients that undergo endoscopic sinus surgery must routinely complete nasal irrigations to maintain the patency of the sinuses and to encourage healing. The current standard of treatment is saline irrigations. Manuka honey has already shown promise in the field of wound healing. The Manuka Honey will be used as the treatment arm in this study and will be compared to the current standard of care, the saline irrigations.

Once the subjects have signed the consent form, they will undergo endoscopic sinus surgery as planned. Randomization (using sealed envelopes) will occur immediately after surgery where patient will receive either the Honey rinse or Saline rinse. There will be 50 envelopes containing a sheet of paper stating "Manuka Honey Irrigation" and another 50 envelopes containing a sheet of paper stating "Saline Irrigation." These envelopes will be sealed, marked with "Nasal Irrigation Study" on the front of the envelope, and mixed in a random fashion. Immediately after surgery, one of these envelopes will be selected to randomize the patient to either the Manuka Honey or Saline irrigation arms. As this is a single-blinded study, the patients will know to which arm they are assigned to, while the primary investigator is blinded.

The standard treatment, as described involves nasal irrigation using a saline solution. This will constitute one arm of the study. The treatment arm will involve the use of the pasteurized Manuka honey nasal irrigation, which is not currently the standard of practice, but is approved by Health Canada to be used for this indication. The subject will use 30cc of the nasal irrigation (to which they are randomized) in each nostril twice daily (once in am, once in pm). No other specific manipulations will be used. The SNOT-22 questionnaire will be administered before the patient is assessed by the clinic physician at 6 days, 5 weeks, and 3 months post-operatively. Patients will not be blinded to the irrigation they are assigned to. The investigators will not know to which arm the subjects have been assigned to.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent.
* Adult (over 19 years of age) patients undergoing sinus surgery for chronic rhinosinusitis (CRS) or allergic fungal sinusitis (AFS).

Exclusion Criteria:

* Co-morbidities, eg. Hypertension, Cardiac Disease, Coagulopathy, CF, Sampter's triad, Diabetes, liver failure
* Medication, eg. Anticoagulants, statins, anti-hypertensives
* Allergies to honey, bee stings

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Post-operative endoscopic appearance | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.
Post-Operative SNOT-22 | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.
  Sino-Nasal Outcome Test (SNOT-22) is current standard in Rhinology for the assessment of the patient's subjective sinus symptoms and its effect on their daily functioning. It is composed of 22 questions, which ask patients to rate their symptoms on a scale of 0-5 (0=no problem, 5=problem as bad as it can be). Questions include patients perceived nasal congestion/blockage, facial pain, fatigue, sadness, etc. This questionnaire is used as the gold standard for patients to rate their subjective symptoms.

SECONDARY OUTCOMES:
Post-operative bleeding | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.
Post-operative pain | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD, FRCSC, Principal Investigator — St. Paul's Hospital, Canada
Locations (1):
- ENT Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Cooper R. Using honey to inhibit wound pathogens. Nurs Times. 2008 Jan 22-28;104(3):46, 48-9. PMID 18293880
- [Result] English HK, Pack AR, Molan PC. The effects of manuka honey on plaque and gingivitis: a pilot study. J Int Acad Periodontol. 2004 Apr;6(2):63-7. PMID 15125017
- [Result] Armstrong DG. Manuka honey improved wound healing in patients with sloughy venous leg ulcers. Evid Based Med. 2009 Oct;14(5):148. doi: 10.1136/ebm.14.5.148. No abstract available. PMID 19794023
- [Result] Alandejani T, Marsan J, Ferris W, Slinger R, Chan F. Effectiveness of honey on Staphylococcus aureus and Pseudomonas aeruginosa biofilms. Otolaryngol Head Neck Surg. 2009 Jul;141(1):114-8. doi: 10.1016/j.otohns.2009.01.005. Epub 2009 Mar 9. PMID 19559969